CLINICAL TRIAL: NCT06043882
Title: Number of Participants Diagnosed With Sarcoidosis by Bronchoscopic Transbronchial Needle Aspiration After Corona Virus Disease of 2019 Infection.
Brief Title: Number of Participants Diagnosed With Sarcoidosis by Bronchoscopic Transbronchial Needle Aspiration After COVID- 2019 .
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU-R 151/2022
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Sarcoidosis; COVID-19
Keywords: Sarcoidosis; COVID-19; SARS-CoV-2; Granulomatous disease
MeSH Terms: conditions — Sarcoidosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the relation between COVID-19 infection and the development of sarcoidosis .: All patients were subjected to the following : history taking , clinical examination , radiological assessment by CT chest , fiberoptic bronchoscopy where biopsies were taken either by conventional TBNA (c-TBNA) , EBUS-TBNA or direct forceps biopsies and sent for histopathological examination and if the patient had past history of COVID-19 infection with previous positive RT-PCR.
  Interventions: Procedure: flexible bronchoscopy

INTERVENTIONS:
Procedure: flexible bronchoscopy — fiberoptic bronchoscopy was done where biopsies were taken either by conventional TBNA (c-TBNA) , EBUS-TBNA or direct forceps biopsies and sent for histopathological examination

SUMMARY:
The goal of this observational study is to learn about sarcoidosis development after COVID-19 infection.

The main question it aims to answer is:

* prevalence of Sarcoidosis among patients previously infected with COVID-19.

Participants will:

* provide previous positive RT-PCR for COVID-19
* Have computed tomography of the Chest with suggestive findings of sarcoidosis
* Have bronchoscopic guided biopsies and pathological analysis to detect number of patients with sarcoidosis.

DETAILED DESCRIPTION:
This prospective cross sectional study was performed on a total of 55 patients with mediastinal and /or hilar lymphadenopathy with or without lung infiltrates referred to Bronchoscopy unit , Chest department, Ain-Shams University hospital for biopsy taking and diagnosis.

All patients were subjected to the following : history taking , clinical examination , radiological assessment by computed tomography (CT )chest , fiberoptic bronchoscopy where biopsies were taken either by conventional-Trans-bronchial needle aspiration (c-TBNA) , endo-bronchial ultrasound (EBUS-TBNA) or direct forceps biopsies and sent for histopathological examination and if the patient had past history of COVID-19 infection with previous positive reverse transcriptase- polymerase chain reaction assay (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with previous positive RT-PCR for COVID -19 and CT chest findings of mediastinal and or hilar lymphadenopathy with or without lung infiltrate will be included. .

Exclusion Criteria:

* Patients younger than 18 years old Patients
* Patients refuse to participate in the study
* Patients previously diagnosed as sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously diagnosed as COVID -19 by RT-PCR ,with mediastinal or hilar lymphadenopathy with or without lung infiltrates referred to bronchoscopy unit ,Chest Department, Ain-Shams University Hospital for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Number and risk factors of sarcoidosis development after COVID -19 infection as diagnosed by TBNA guided tissue biopsies in bronchoscopy unit, chest department, Ain Shams university. | 6 months
  Number of COVID-19 patients diagnosed by TBNA guided biopsies as having granulomatous tissue suggesting sarcoidosis development, and risk factors that associate its development.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda A Mohamed, MD, Principal Investigator — faculty of medicine, Ain Shams university
Locations (1):
- Hoda atiatullah, Cairo, Egypt